CLINICAL TRIAL: NCT06942455
Title: A Sleep Hygiene Intervention to Improve Sleep Health in Urban, Latino Middle School Children
Acronym: SIESTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MD019452 (NIH); R01MD019452 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-24 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Sleep Quality; Intervention Study; Ethnic Minority
Keywords: pediatric sleep intervention; sleep hygiene intervention; intervention determinants; sleep outcomes
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The primary aim of this study is to test the SIESTA intervention through a large-scale Randomized Control Trial. 300 Latino middle school aged youth (11-13 years old, grades 6-8) will be randomly assigned either to the SIESTA intervention, or to the Sleep Education plus Child Health attention-control condition. Treatment effects on primary (e.g., sleep duration, sleep efficiency) and secondary (e.g., sleep hygiene) outcomes will be evaluated. Assessments will occur at a baseline visit and immediately following the conclusion of the intervention, and at 4, 8, and 12 months after the intervention.
Masking Description: The research assistants collecting outcomes data post-intervention will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIESTA (Experimental): The SIESTA Intervention includes 4, 60-minute group remote sessions by a trained facilitator, and 2, 90-minute family sessions in their home 1 week after group Sessions 1 and 4. SIESTA incorporates key sleep hygiene principles and strategies critical to optimal sleep health in middle schoolers and tailored to urban Latino children's cultural background and urban setting. Areas of focus include the importance of adequate sleep duration, principles and strategies to enhance sleep hygiene, and characteristics of healthy sleep environments, and were developed with targeted goals. After intervention group Session 1, daily sleep questions about the child participant are completed, including key sleep parameters (bedtime, rise time, night awakenings) and sleep hygiene behaviors (daytime naps, electronics, caffeine use) via Qualtrics. Responses are summarized and presented pictorially in caregiver-child sessions to facilitate developing sleep goals for the youth and assess their progress.
  Interventions: Behavioral: SIESTA
- Sleep Education plus Child Health attention control (Other): A facilitator from the community will deliver this attention control condition, which consists of the same number of sessions as SIESTA but will focus only on basic sleep hygiene education plus general child health topics (e.g., nutrition, physical activity, safety). It is expected that this will exert limited treatment effects on sleep hygiene, because it does not 1) involve effective behavioral approaches for this age group, or 2) include content tailored for urban Latinos.
  Interventions: Behavioral: Sleep education and health education control

INTERVENTIONS:
Behavioral: SIESTA — Active condition
  Arms: SIESTA
Behavioral: Sleep education and health education control — Attention Control
  Arms: Sleep Education plus Child Health attention control

SUMMARY:
The main goal of this study is to evaluate the "SIESTA" intervention, a culturally and contextually tailored sleep hygiene intervention that has the potential to exert greater improvements in sleep hygiene and sleep outcomes for group that may be more vulnerable to poor sleep health.

The main question is: do SIESTA participants have improved sleep outcomes, sleep hygiene behaviors and less sleep-related impairment compared to Control Group participants?

Participants randomized to the SIESTA intervention will:

1. Attend 4 remotely administered group sleep hygiene education sessions
2. Complete along with a parent/guardian, two individualized sessions administered by a SIESTA intervention facilitator
3. Complete study survey at baseline, end of treatment, and at 4, 8 and 12 months post-intervention.
4. Wear electronic sleep watches (actigraphy) throughout the protocol to objectively measure sleep duration and quality.

Participants randomized to the Child Health Control condition will:

1. Attend 4 remotely administered group sessions covering general health topics
2. Complete along with a parent/guardian, two individualized sessions administered by a SIESTA intervention facilitator
3. Complete study survey at baseline, end of treatment, and at 4, 8 and 12 months post-intervention.
4. Wear electronic sleep watches (actigraphy) throughout the protocol to objectively measure sleep duration and quality.

A secondary goal of the study is to conduct a process evaluation to prepare for future larger scale use of the intervention in other urban school settings. This will entail assessing Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) of the program through several methods, such as by conducting in-depth interviews with research participants and their parents/guardians, as well as school staff and by looking at rates of participation in the program.

DETAILED DESCRIPTION:
Sleep is essential for optimal health and development. Poor sleep is associated with impaired functioning and academic performance, and worse health outcomes in children. Latino children are disproportionately present in urban settings, and due to their exposure to higher levels of urban and cultural stressors, are at greater risk for poor sleep hygiene and quality.

SIESTA (School Intervention to Enhance Latino Students' Time Asleep) is a novel sleep hygiene intervention for improving sleep hygiene and sleep duration in urban Latino middle schoolers in two geographic areas with a high proportion of urban Latino children at increased risk for poor sleep health: Providence, Rhode Island, and San Juan, Puerto Rico.

SIESTA involves 4 group sessions administered in school to Latino middle schoolers (6th-8th grade) and two child-caregiver sessions administered remotely by a bilingual (English/Spanish) trained facilitator from the community.

The goal of this project is to administer a two-site hybrid type 1 effectiveness-implementation design to evaluate SIESTA's effects on a larger-scale- for addressing Latino middle schooler's sleep health, while also assessing implementation determinants.

The first aim of the study is to evaluate SIESTA through a large-scale RCT with urban middle school students in Providence, RI and San Juan, Puerto Rico. The researchers will enroll 150 Latino children per site (N=300), and randomly assign them either to the SIESTA intervention, or to the Sleep Education plus Child Health attention-control condition (9 groups of each of the two conditions, per site; 8-9 students per group). Treatment effects on primary sleep outcomes will be evaluated, including sleep duration, efficiency and sleep onset latency. Secondary sleep outcomes will include sleep hygiene behaviors, the sleep environment, and sleep-related disturbances and impairment. Assessments will occur prior to, immediately following, and at 4, 8, and 12 months after the intervention.

Each participant will be active in the protocol over approximately 14 months, during which it is hypothesized that SIESTA participants will have improved sleep outcomes, sleep hygiene behaviors and less sleep-related impairment relative to Controls.

The second study aim is to identify implementation determinants and preliminary implementation outcomes of SIESTA to prepare for future large-scale implementation in other urban school settings. A mixed methods process evaluation will be implemented, with input from community partners using the RE-AIM framework throughout and following administration of the RCT.

SIESTA has the potential to improve sleep outcomes in urban Latino children and their daytime functioning, and to address a critical gap of the need for tailored and effective sleep hygiene interventions for children at greater risk for poor sleep health.

ELIGIBILITY:
Inclusion Criteria:

* children must be middle schoolers between 11-13 years old, live and go to school in one of the targeted school districts and sleep no more than 9 hours on an average night

Exclusion Criteria:

* Children are not eligible to take part in the study if they have a medical, psychiatric, or developmental condition and/or are taking medicine for any condition that might affect their ability to and comfort with taking part in the study.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Duration | Sleep duration will be assessed for 1-2 weeks at baseline, immediately after the intervention ("end of treatment") and at follow ups at 4, 8, and 12 months post intervention/control.
  Sleep Duration through actigraphy will be calculated through Time in Bed (TIB) scores. A daily diary will document sleep events (e.g., bedtime) to score actigraphic data . Children will wear the actigraph Motion Logger device for 1-2 weeks at each time point. Data will be compared to data in a family-report daily diary using standard procedures.
Sleep Efficiency/Quality | Sleep efficiency will be assessed for 1-2 weeks at baseline, end of treatment and at each 4, 8, and 12 months post intervention/control.
  Sleep efficiency will be estimated via actigraphy and will be calculated through % epochs of sleep between sleep start and sleep end.

SECONDARY OUTCOMES:
Sleep Disturbance and Sleep-related Impairment | Sleep Disturbance and Sleep-related Impairment measures will be collected on each child at each of the of the 5 research assessment time points: enrollment/baseline, immediately after the intervention, and at the 4, 8 and 12 month follow up visits.
  Sleep disturbance and sleep-related impairment will be assessed by caregiver and child report by the Patient-Reported Outcomes Measurement Information System (PROMIS™) measures (Yu et al., 2011). Participants will be asked to report on the previous week. Raw scores are converted to T-scores (Mean=50, SD=10). Higher scores indicate more of the concept being measured, hence higher scores on Sleep Disturbance and Sleep Impairment indicate less optimal status on these domains, while scores lower than T=50 indicate better functioning (less sleep disturbance and sleep impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Koinis-Mitchell, PhD, Principal Investigator — Alpert Medical School of Brown University; Ligia Chavez, PhD, Principal Investigator — University of Puerto Rico Medical Sciences Campus
Locations (2):
- Rhode Island Hospital, Providence, Rhode Island, United States
- Centro Medico, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
The final datasets will include individual participant survey data, diary data, and aggregated daily-level actigraphy data. We will share cleaned and de-identified individual-participant level data where all HIPAA identifiers have been removed. The rationale for sharing only cleaned data is to facilitate data reuse. All data will be made available through a user agreement.
  A README file and data dictionary will be generated and deposited into a repository along with all shared datasets. Documentation will include a description of the study design and methods, survey measures, data acquisition devices (actigraphy), and any other tools (e.g., software, databases, services) used in the study or in processing the data. The data dictionary will describe all variables in the dataset. The finalized SIESTA and Control Group Training manuals for group facilitators, and the SIESTA and Control Group Intervention manuals will be available in English and Spanish.
Supporting Information: Study Protocol
Time Frame: Outcomes data related to the primary specific aims will be available at the time of publication; all other generated data will be shared when data processing is complete. All study data will be stored in the repository for at least 5 years.
Access Criteria: The National Sleep Research Resource (NSRR) funded by NHLBI is a potentially suitable repository. The MPIs will review this and other options during study implementation and will consult the data management experts at their institution and collaborators with relevant expertise. The final decision for repository will be made by the MPIs with consultation on best practices for data preservation for this study from these resources/ colleagues.